CLINICAL TRIAL: NCT06676982
Title: Clinical Trial of Autologous CD19 CAR-T Cells (CNCT19) Therapy for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001017
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Advanced Hepatocellular Carcinoma; CAR-T; CD19; Tumor-associated macrophage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): CNCT19
  Interventions: Biological: anti-CD19 CAR-T

INTERVENTIONS:
Biological: anti-CD19 CAR-T — All subjects were intravenous administrated with CNCT19 CAR-T.

SUMMARY:
A phase I clinical study of the safety and tolerability, efficacy of CNCT19 CAR T-cell therapy in patients with advanced hepatocellular carcinoma hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a single-arm, dose-escalation, open, exploratory clinical study to evaluate the safety and tolerability, preliminary efficacy and PK/PD haracteristics of CNCT19 CAR T-cell therapy in the treatment of advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years, male or female;
* Subjects voluntarily participated in the research and signed the Informed Consent Form (ICF) by themselves or their guardians;
* Pathologically diagnosed with hepatocellular carcinoma, patients with China liver Cancer Staging (CNLC) stageII-III.;
* HCC patients who are not suitable for surgical resection or local treatment (including ablation therapy, interventional therapy, and radiation therapy), or who experience recurrence or progression after surgery and/or local treatment, and who have previously received at least second-line systematic standardized treatment and have progressed or are intolerant to it;
* According to RECIST 1.1 standard, there should be at least one measurable tumor lesion;
* Tumor samples that meet the requirements (paraffin blocks or unstained sections with a quantity that meets the testing requirements specified in this study) within 2 years, and have CD19/CD68 double positive cells detected by immunohistochemistry or immunofluorescence;
* Child-Pugh ≤ 7 and no history of hepatic encephalopathy;
* ECOG 0-1;
* Expected survival period ≥ 12 weeks;
* The toxicity caused by previous treatment has stabilized or recovered to ≤ level 1 (except for cases judged by the researcher to be clinically insignificant)

Exclusion Criteria:

* Active brain metastasis;
* Patients who have received or are waiting for organ transplantation;
* Active autoimmune diseases that require systemic immunosuppressive therapy within the past 2 years, such as systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis, etc;
* Researchers evaluated that the proportion of intrahepatic tumors is greater than 50% of the entire liver; Or there may be tumor thrombus formation in the main portal vein, or tumor thrombus invasion into the mesenteric vein/inferior vena cava;
* Use any of the following drugs or treatment methods within the specified time before cell collection: a Received local treatments such as surgical intervention, radiation therapy, ablation, etc. for the studied disease within 4 weeks prior to cell collection; b. Patients who have undergone major surgical procedures or significant trauma within 4 weeks prior to cell collection, or who are expected to undergo major surgery during the study period; c. Received immunotherapy such as anti-PD-1 and PD-L1 within one week prior to cell collection; d. Received chemotherapy drugs or targeted therapy such as sorafenib, regorafenib, lenvatinib within 2 weeks prior to cell collection; e. Used therapeutic doses of corticosteroids within 3 days prior to cell collection, but allowed to use topical and inhaled corticosteroids;
* Within the past 5 years or simultaneously with other incurable malignant tumors, except for cervical cancer in situ, basal cell carcinoma of the skin, and ductal carcinoma in situ of the breast;
* Individuals who have received other cell therapies or gene modified cell therapies in the past;
* Central nervous system diseases that have clinical significance in the past or screening, such as epilepsy, epileptic seizures, cerebrovascular disease (ischemia/hemorrhage/cerebral infarction), cerebral edema, reversible posterior white matter encephalopathy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome or psychiatric disorders;
* There are chronic obstructive pulmonary disease, interstitial lung disease, and clinically significant abnormalities in lung function tests;
* After evaluation by the researchers, it was found that the subject had a large amount of uncontrollable serous fluid accumulation (such as pleural effusion, abdominal effusion, pericardial effusion).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Within 28 days of CNCT19infusion
  Describe the adverse events of limiting further increases in the dose of CNCT19.
Adverse events | Within 24 months after the treatment
  Describe adverse events (AEs) and serious adverse events (SAEs) that are "likely" or "definitely" related to the studytreatment that occur at any time of 24 months after treatment.
Maximum tolerated dose | From enrollment of the first subject to completion of follow-up of the last subject (up to 3 years)
  Determine the optimal agent for CNCT19 at maximum tolerated dose.

SECONDARY OUTCOMES:
Effectiveness evaluation | From treatment of the first subject to completion of follow-up of the last subject (up to 3 years)
  Objective response rate by RECIST 1.1.
Effectiveness evaluation | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  Progression-free survival by RECIST 1.1
Effectiveness evaluation | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  Duration of response by RECIST 1.1
Effectiveness evaluation | From enrollment of the first subject to completion of follow-up of the last subject (up to 3 years)
  Time to response by RECIST 1.1
Effectiveness evaluation | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  Disease control time by RECIST 1.1
Pharmacokinetic evaluation | Within 28 days of CNCT19 infusion
  Detect duration of CAR-T cells in vivo.
Pharmacokinetic evaluation | Within 28 days of CNCT19 infusion
  Detect expansion of CAR-T cells in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Professor, Principal Investigator — Zhejiang University
Locations (2):
- China (2):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - First Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No